CLINICAL TRIAL: NCT05717985
Title: A Randomized Controlled Trial to Compare De-epithelized Connective Tissue Grafts and Modified Combined Approach for Connective Tissue Grafts
Brief Title: Evaluation of De-epithelized Connective Tissue Grafts and Modified Combined Approach for Connective Tissue Grafts
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: GGPM-2022-024
Record Dates: First submitted 2023-01-17; First posted 2023-02-08 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Gingival Recession
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- de-epithelized gingival graft (Active Comparator): A type of mucogingival surgery where a gingival graft is harvested from the palate, prepared chairside and placed on a recipient site to augment it. Dressing material and sutures is placed at the donor site.
  Interventions: Procedure: de-epithelized gingival graft
- modified combined approach (Experimental): A type of mucogingival surgery where a gingival graft is harvested from the palate, prepared chairside and placed on a recipient site to augment it. A part of the prepared tissues namely the epithelial layer is replaced at the donor site and sutured.
  Interventions: Procedure: modified combined approach

INTERVENTIONS:
Procedure: modified combined approach — A thin layer of epithelium will be excised from the harvested graft. This epithelium will be replaced at the donor site and sutured.
  Arms: modified combined approach
Procedure: de-epithelized gingival graft — Only dressing material will be placed at the donor site after graft harvesting
  Arms: de-epithelized gingival graft

SUMMARY:
This study aims to compare the de-epithelized gingival graft (control group) and modified combined approach for connective tissue graft (test group) in patients undergoing palatal graft harvesting for mucogingival surgery in the oral cavity

DETAILED DESCRIPTION:
Harvesting a palatal mucosal tissue graft as an autologous donor for oral soft tissue augmentation is widely practiced. Tissue harvest in patients with anatomically thin phenotypes can cause significant morbidity and compromised healing process. The modified combined approach (MCA) for connective tissue grafts has the potential for faster healing and fewer postoperative complications, compared to the recommended harvesting technique of de-epithelized gingival graft (DGG). However, the modified combined approach for connective tissue grafts have yet to be extensively investigated.

This examiner-masked, randomized study aims to compare post-operative morbidity and treatment outcomes in patients undergoing modified combined approach for connective tissue graft (test group) compared to the de-epithelized gingival graft (control group) harvesting techniques in tissue augmentation.

Participants will be randomized into two groups receiving one of either modified combined approach for connective tissue graft or de-epithelized gingival graft. Collection of the study parameters will utilize both examiner-assessed, and patient reported outcomes.

The study will report on the optimum palatal mucosal graft harvesting technique in an Asian population. The findings of this study will be utilized to formulate clinical recommendations for soft tissues augmentation in this population.

ELIGIBILITY:
Inclusion Criteria

* systemically healthy subjects;
* able to give informed consent;
* age ≥ 18 years;
* requiring palatal tissue harvesting for soft tissue augmentation in the oral cavity

Exclusion Criteria:

* subjects with periodontal diseases;
* subjects with poor oral hygiene of >30% plaque index;
* pregnant or lactating females;
* subjects taking medication with any known effect on the periodontal soft tissues;
* subjects with pathology in the oral cavity causing any degree of pain;
* subjects wearing removable or fixed prothesis that is in contact with the donor site an
* those with allergies to painkillers including ibuprofen and paracetamol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-02-22 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Pain after gingival graft harvesting | up to 3 months after surgery
  Measured using a self-reported questionnaire that is designed by the research group. The pain will be measured using a visual analogue score (minimum value=0 and maximum value=10), and using a surrogate measure of amount of painkillers taken by the participants after the surgery (minimum value= 0, maximum value= 2 grams for paracetamol, 1200 mg for ibuprofen). Higher score on the visual analogue scale and higher amount of painkillers taken is a worst outcome.

SECONDARY OUTCOMES:
Healing after gingival graft harvesting | up to 3 months after surgery
  Measured clinically by the investigators. The donor site will be inspected and scored using the Wound Healing Index (Landry et. al, 1988). The photograph of the donor site will also be taken and analysed digitally to measure the amount of keratinisation using the ImageJ Software. Higher score on the Wound Healing Index is a better outcome (minimum score= 0, maximum score= 5). Higher amount of keratinised tissue as measured by the software is a better outcome (minimum value= 0, maximum value= the full surface of the donor site estimated at 3200 square mm).

CONTACTS AND LOCATIONS:
Overall Officials: Nik Madihah Nik Azis, DClinDent, Study Director — Faculty of Dentistry, University Kebangsaan Malaysia
Locations (1):
- Faculty of Dentistry, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No